CLINICAL TRIAL: NCT04174911
Title: A Randomized Phase 2a, Double-blind, Placebo-Controlled Study Examining the Safety and Efficacy of BOL-DP-o-08 in Patients With Endometriosis Syndrome.
Brief Title: A Study to Evaluate the Safety and Efficacy of BOL-DP-o-08 in Patients With Endometriosis Syndrome.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: covid 19
Sponsor: Breath of Life International Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOL-P-09
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOL-DP-o-08 (Experimental): BOL-DP-o-08
  Interventions: Drug: BOL-DP-o-08
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOL-DP-o-08 — BOL-DP-o-08 sublingual drops
  Arms: BOL-DP-o-08
Drug: Placebo — sublingual drops
  Arms: Placebo

SUMMARY:
A Phase 2a, Single-center, randomized, double-blind, placebo-controlled study, in 80 subjects diagnosed with Endometriosis, stage 2-4

DETAILED DESCRIPTION:
Subjects diagnosed with Endometriosis will be eligible for enrollment. During a Screening Period of 2 weeks, inclusion and exclusion criteria will be assessed to determine if they are eligible to move into the Treatment Period.

During Treatment, subjects will randomly receive either BOL-DP-o-08 or placebo TID for 16 weeks. At the end of the treatment, a follow-up visit for safety assessments will be conducted 4 weeks after the termination visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, aged 18 years old
* Regular menstrual cycles
* Endometriosis diagnosed by ultrasonography and gynecological examination, or laparotomy, laparoscopy or imaging analysis (combination of magnetic resonance imaging and ultrasonography) of endometriotic ovarian chocolate cysts
* The presence of subjective symptoms during menstruation (at least one from among lower abdominal pain, lumbago, defecation pain, nausea and headache
* The presence of subjective symptoms during non-menstruation (at least one from among lower abdominal pain, lumbago, defecation pain, dyspareunia, and pain on internal examination)
* The presence of objective findings (induration in the pouch of Douglas and/or limited uterine mobility).
* Subject is on stable therapy regimen for at least 8 weeks prior to screening period
* Subjects able and willing to comply with the requirements of the protocol
* Subjects able to understand and sign written informed consent to participate in the study

Exclusion Criteria

* Undiagnosed genital bleeding
* Class 3 or more pap test within 3 months before enrollment
* Use of GnRH agonist, testosterone derivatives, hormonal therapy with progesterone and/or estrogen, estrogen antagonists or aromatase inhibitors within 16 weeks before enrollment
* Having undergone surgery therapy or surgical examination for endometriosis within menstrual cycle before the start of medication
* Use of drugs that could be expected to affect the release of sex hormones (e.g. sulpiride, cimetidine)
* A history or complication or finding of thrombosis/embolism or depression
* Malignant tumor complication or finding suggestive of a malignant tumor
* Complication of serious heart, liver, kidney, blood or endocrine disease
* Participation in another clinical trial within 4 months before enrollment
* Patients deemed unsuitable for study entry by the investigator
* Subject with other severe pain due to other conditions that may confound assessment or self-evaluation of the pain associated with endometriosis
* Subject with serious cardiovascular, hepatic, renal, respiratory, gastrointestinal, urological, neurological, endocrine, autoimmune or hematological disease, malignancy not considered cured (except for BCC) or clinically significant laboratory or electrocardiogram abnormality which indicate a serious medical problem or require significant intervention in the judgment of the investigator
* Current systemic infection
* Subject with a diagnosis of social phobia, generalized anxiety disorder, bipolar disorder, psychosis, major depressive disorder or schizoaffective disorder; or any other disorder with psychotic symptoms - based on the clinical opinion of the investigator.
* Subject with personality disorder or mental retardation
* Subjects with known allergy to one or more of the study drug components
* Female subject who is pregnant, lactating, or who want to get pregnant during the study period
* Female of child-bearing potential who can't agree to utilize medically acceptable and reliable means of birth control during the study and for 1 month following the last dose of the study
* Subject with a history of alcohol or any psychoactive substance abuse or dependence (including alcohol, but excluding nicotine and caffeine) within the past 1 year
* Subject receiving opiates or cannabis therapy
* Patients with first degree siblings with significant mental or psychiatric disorder or a psychiatric disease (especially patients less than 30 years old)
* Subject who are using one of the following medications: Opiates, Primidone, Phenobarbitol, Carbamazepine, Rifampicin, Rifabutin, Troglitazone and Hypericum perforatum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in a pain Numeric Rating Scale | Baseline to week 16
  The Visual Analogue Scale (VAS) is a Numeric Rating Scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers)

SECONDARY OUTCOMES:
Change in Clinical Global Impression | Baseline to week 16
  Clinical Global Impression is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (among the most severely ill patients)
Changes in the size of endometrial ovarian cysts and endometrial nodules | Baseline to week 16
  measured by gynecological Ultrasound examination

IPD SHARING:
Plan to Share IPD: No